CLINICAL TRIAL: NCT00817271
Title: A Randomised, Open, Two-Way Cross-Over, Phase I Study to Evaluate the Response to Glucagon Versus the Spontaneous Counter-Regulatory Response in T2DM Patients Treated With AZD1656 and Metformin During Hypoglycemia
Brief Title: To Evaluate the Response to Glucagon During Hypoglycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00018
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Type 2 Diabetes
Keywords: Type II Diabetes; Counter-regulatory response; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — AZD1656; Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD1656; Drug: Glucagon
- 2 (Experimental)
  Interventions: Drug: AZD1656

INTERVENTIONS:
Drug: AZD1656 — Dose titration of oral suspension during 2 days to a tolerable dose given twice daily. Subjects will thereafter be treated with this dose for another 6 days. On day 5 and 8 the dose will be given as a single dose
Drug: Glucagon — 1 mg injected 3 hr post AZD1656 morning dose on day 5 alt. day 8
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the response to Glucagon versus the spontaneous hormonal response to low blood sugar levels in T2DM Patients treated with AZD1656 and Metformin

ELIGIBILITY:
Inclusion Criteria:

* type II diabetes patients, female with non child-bearing potential
* T2DM diagnosis confirmed by C-peptide >0.3nmol/L and no glutamic acid decarboxylate (GAD) antibodies at enrolment (screening)
* Treatment with metformin alone with a total daily dose not less than 1 000 mg. Stable glycaemic control indicated by unchanged treatment within 3 months prior to enrolment

Exclusion Criteria:

* History of ischemic heart disease, symptomatic heart failure, stroke, transitory ischemic attack or symptomatic peripheral vascular disease
* Signs of diabetic proliferative retinopathy or diabetic maculopathy, at screening or on an ophthalmological examination within 3 months from start of study
* Participating in another clinical study during the last 30 days prior to enrolment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
P-Glucose levels | Repeated sampling during the 24 hour period on day 5 and 8

SECONDARY OUTCOMES:
Safety and tolerability (AE, BP, pulse, plasma glucose, laboratory variables, weight and ECG) | Frequent measurements during the study period
Pharmacokinetic variables (Area under the plasma conc-time curve from time 0 to 24 hours post dose (AUC0-24), maximum plasma conc(Cmax), time to reach maximum plasma conc(tmax), terminal elimination half-life and apparent oral clearance | Repeated sampling during the 24 hour period on day 5 and 8
Pharmacodynamics (P-Glucose, S-Insulin and S-C-peptide) | Repeated sampling during the 24 hour period on day 5 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof., Study Director — AstraZeneca R&D Mölndal; Marcus Hompesch, MD, Principal Investigator — Profil Institut for Clinical Research Inc.
Locations (1):
- Research Site, Chula Vista, California, United States